CLINICAL TRIAL: NCT06161246
Title: An Open-label, Randomized, Split-face, Controlled Study on Pain Management With Injection of Botulinum Toxin for Glabellar Line Correction
Brief Title: A Controlled Study on Pain Management With Injection of Botulinum Toxin for Glabellar Line Correction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Collaborators: DeNova Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.US.SL.028
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-10

CONDITIONS: Injection Site Discomfort

STUDY DESIGN:
Intervention Model Description: Subjects will receive comfort intervention on one side of face, and will not receive comfort intervention on the other side of face.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Group (Experimental): Subjects will be treated for correction of glabellar lines with Dysport and comfort intervention on one side and Dysport only on the other side depending on pre-determined randomization. Subjects will complete the study assessments and end the study.
  Interventions: Device: Vibrating Beauty Bar

INTERVENTIONS:
Device: Vibrating Beauty Bar — A vibrating beauty bar will be used at the injection site for patient comfort.
  Other Names: Vibration therapy

SUMMARY:
This is an open-label, single-center, randomized, split-face, controlled study to assess the effect of comfort intervention on pain during treatment injection compared against non-comfort intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects aged 18-65 years
* Females or males
* Having any Fitzpatrick skin types I-VI
* Any races and ethnicities
* Having any self-assessed pain tolerance, with a minimum of 5 subjects in each category (low, medium, and high pain tolerance)
* Subject with intent to undergo correction of the glabellar lines (frown lines between the eyebrows)
* Subject with moderate-to-severe glabellar lines as assessed by investigator using Glabellar Line Severity Scale (GLSS).
* Subject with no history of aesthetic injection, i.e., botulinum toxin, collagen, hyaluronic acid, calcium hydroxyapatite, poly L-lactic acid or permanent materials.
* Subject with healthy immune systems
* Subject willing to abstain from any other facial plastic surgical or cosmetic procedure(s) during the duration of the study.
* For female subjects of childbearing potential, she must not be pregnant, breastfeeding or planning pregnancy during the course of the study. Subjects must be willing to take a urine pregnancy test (UPT) prior to all treatment injections.
* Ability of giving consent for participation in the study
* Agreement to adhere to the procedures and requirements of the study and to report to the site on the day(s) and at the time(s) scheduled for the assessments

Exclusion Criteria:

* Pregnant, breastfeeding, or planning pregnancy during the course of the study, confirmed by UPT.
* Current smokers or consumer nicotine (e.g., cigarettes, e-cigarettes, vaping device with pre-filled pods, vapor tank or mod, chewing tobacco)
* History of allergy or hypersensitivity to botulinum toxin type A, human albumin, lactose, or cow's milk protein
* Subject with signs and symptoms of eyelid or brow ptosis, inability to substantially lessen glabellar lines by physically spreading them apart, or history or presence of facial nerve palsy, as judged by the Investigator.
* Previous or present multiple allergies or severe allergies, such as manifested by anaphylaxis or angioedema, or family history of these conditions.
* Previous aesthetic treatment in the face with any of the following injection prior to the baseline visit:

  1. Botulinum toxin
  2. Collagen, hyaluronic acid
  3. Calcium hydroxylapatite, poly L-lactic acid, fat or permanent materials (non-biodegradable)
* Previous treatment/procedure in the face in the previous 2-4 weeks that, in the Investigator's opinion, would interfere with the study injections and/or study assessments or exposed the study subject to undue risk by study participation, or planning to undergo any of these procedures affecting the treatment area at any time during the study e.g.,

  1. Resurfacing (laser, photo modulation, light, radiofrequency, ultrasound, chemical peel, dermabrasion, or other ablative/non-ablative procedures)
  2. Needling or mesotherapy
  3. Cryotherapy
* Presence of any disease or lesions near or on the glabellar region, e.g.,

  1. Inflammation, active, or chronic infection in or near the treatment area
  2. Psoriasis, eczema, rosacea, atopic dermatitis, herpes zoster/herpes simplex, and acanthosis
  3. Scars or deformities
* History of bleeding disorders or treatment with anticoagulants or inhibitors of platelet aggregation (e.g., aspirin or other non-steroidal anti-inflammatory drugs), omega 3, or vitamin E within 14 days before treatment. Omega 3 and vitamin E are acceptable only as part of a standard multivitamin formulation.
* Planning on having surgeries and/or invasive medical procedures during the course of the study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Baseline
  Visual Analogue Scale is a 11-point psychometric scale that specifies the level of pain. Subject will be shown a photo of a VAS and verbally report a pain score between 0 and 10, which will be captured by a clinic staff. A score of 0 corresponds to no pain felt and a score of 10 corresponds to very high pain.

SECONDARY OUTCOMES:
Self-assessment questionnaire | Baseline
  To evaluate investigator and subject's satisfaction and preference on treatment experience using self-assessment questionnaires on treatment injection with and without comfort intervention

CONTACTS AND LOCATIONS:
Locations (1):
- DeNova Research, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No